CLINICAL TRIAL: NCT04064775
Title: The Influence of Fictitious Peers in a Social Media Intervention for Downsizing Portions: The Smart Snacking Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Leeds (Other)
Collaborators: Coventry University (Other); Penn State University (Other)
Responsible Party: Principal Investigator, Charlotte Evans, Principal investigator, University of Leeds
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17-0111/ 17-0094
Record Dates: First submitted 2019-05-16; First posted 2019-08-22 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Eating Behavior; Social Psychology
Keywords: Social influence; Peer influence
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Intervention 2 used a parallel design where participants were either allocated to an intervention or a control group in a between-subjects repeated measures design.
Who Masked: Participant
Masking Description: Participants were informed they were in a study about snacking behaviour but were not told that we were attempting to reduce their portion sizes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smart snacking intervention (Experimental): In intervention 2 participants took part in a 4-week intervention on Instagram. Participants saw images of fictitious peers' snacks or beverages three times per week, and saw snack information images three times per week. Peer snack images were posted on days 2,4 and 6 of each week, and snack information images were posted on days 1,3 and 5 of each week. Images were posted between 10-11am each day. Participants also completed quizzes related to snacking at the end of weeks 1-3. Participants completed a survey at baseline and intervention end to assess their ideal portion sizes to allow for examination of the effectiveness of the intervention.
  Interventions: Behavioral: Smart snacking intervention
- Control (No Intervention): Participants in the control received no intervention. They completed the questionnaires at the end of weeks 1, 2 and 3, and also completed the surveys at baseline and intervention end.

INTERVENTIONS:
Behavioral: Smart snacking intervention — The smart snacking intervention aimed to examine whether peer-led nudging on social media influenced adolescents to reduce their self-reported ideal portion sizes for a variety of HED snacks and SSBs. In intervention 2, participants were randomly allocated to the intervention or control condition, and their ideal portion sizes were assessed through a survey at baseline and intervention end.
  Arms: Smart snacking intervention

SUMMARY:
The 2 interventions aimed to examine whether peer-led nudging on social media may be a way of influencing young adults and adolescents to reduce their self-reported ideal portion sizes of high energy-dense snacks and sugar-sweetened beverages.

DETAILED DESCRIPTION:
Two pilot interventions were conducted which examined the influence of peer-led nudging on social media as a way of influencing self-reported ideal portions of high energy-dense snacks and sugar-sweetened beverages. In both interventions the peers posted images of 'their' snacks and beverages, which constituted the recommended portion, onto an Instagram account. The peers also posted images relating to portion sizes, calories and other information related to health but not specifically portion size. It was hypothesised that viewing images of peers' snacks would influence the participants to reduce their own snack and beverage ideal portion sizes.

Intervention 1 lasted for 2 weeks and recruited young adults and used a within-subjects design. Intervention 2 lasted for 4 weeks and recruited adolescents and used a between-subjects design. In intervention 2, participants were randomly assigned to either the intervention or the control condition. This protocol focusses on intervention 2.

In both interventions, participants in the intervention condition were added to an Instagram account and were required to visit Instagram daily and to like all posts. All participants (intervention and control) completed a survey at baseline and at the end of the intervention, and completed quizzes at the end of each week.

ELIGIBILITY:
Inclusion Criteria:

13-16 years old (intervention 2)

Exclusion Criteria:

* Younger than 13 or older than 16 (intervention 2).
* History of or current eating disorder

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Self-reported ideal portion size | Baseline at the beginning of week 1 and intervention end at the end of week 4.
  Questionnaire measuring participants' self-reported ideal portion size. The aim of the intervention was to reduce the ideal portion size. Participants were provided with different images of food. For each image, judgements were made on whether the portion was 'too little', 'slightly less than I would eat', 'just right', 'slightly more than I would eat', or 'too much'.

SECONDARY OUTCOMES:
Perceptions of peers' ideal portion sizes | Baseline at the beginning of week 1 and intervention end at the end of week 4
  Questionnaire measuring participants' perceptions of their peers' ideal portion sizes. Participants were provided with images of different energy dense foods. For each image, judgements were made on whether the portion was 'too little', 'slightly less than I would eat', 'just right', 'slightly more than I would eat', or 'too much'. The aim of the intervention was to reduce the ideal portion size.
Participants liking and frequency of consumption of high energy dense snack foods and sugar-sweetened beverages | Baseline at the beginning of week 1 and intervention end at the end of week 4
  Questionnaire measuring participants' liking and frequency of consumption. Participants' reported frequency of consumption for and liking of each item were assessed based on questions used by Stok, De Ridder, De Vet, & De Wit (2014). Mean frequency and liking scores were calculated for HED snacks and SSBs. A low score for frequency indicated that the item was not eaten frequently, a low score for liking indicated that the item was not liked.
Participants' intentions regarding their portions | Baseline at the beginning of week 1 and intervention end at the end of week 4
  Questionnaire measuring participants' intentions. Participants' reported intentions which were assessed based on questions used by Stok, De Ridder, De Vet, & De Wit (2014). Mean intention scores were calculated for HED snacks and SSBs. A low score for intention score indicated that participants did not intend to change their behaviour.

IPD SHARING:
Plan to Share IPD: No
Data will be available on request. Only anonymised data will be available.